CLINICAL TRIAL: NCT00843622
Title: A Controlled Study of the Ability of a Traditional Swedish Smokeless Tobacco Product ("Snus") to Increase the Quit Rate Among Cigarette Smokers Who Wish to Stop Smoking
Brief Title: Controlled Study of the Ability of a Smokefree Tobacco Product to Increase the Quit Rate Among Cigarette Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Match AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM 08-01
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Cigarette Smoking
Keywords: Smoking; Smoking cessation; Smokeless tobacco; Snus
MeSH Terms: conditions — Cigarette Smoking; Smoking; Smoking Cessation; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tobacco-based, smokefree product in pouch format for oral use, pouch size 1.0 or 0.5 g to be used ad libitum by participants
  Interventions: Drug: Low-nitrosamine smokefree tobacco product for oral use
- 2 (Placebo Comparator): Non-tobacco, non-nicotine placebo product in pouch format for oral use, pouch size 1.0 g or 0.5 g, to be used ad libitum by the participants
  Interventions: Other: Non-tobacco, non-nicotine placebo product

INTERVENTIONS:
Drug: Low-nitrosamine smokefree tobacco product for oral use — Smokeless tobacco in paper sachets containing 1.0 or 0.5 g of the product. Usage ad libitum. Recommended dosages: 10-24 sachets per day (1.0 g sachets). Among participants who typically smoke >15-20 cigarettes per day and/or has a Fagerström score of 7 or higher, the recommended maximum number of sachets per day is 30. For participants who use small sachets (0.5 g) the recommended daily use is double compared that of 1.0 g sachets.
  Other Names: Swedish tobacco-based smokefree product for oral use ("General"-type Swedish "snus"); Placebo "snus" ("Onico"-type product)
  Arms: 1
Other: Non-tobacco, non-nicotine placebo product — Placebo product in paper sachets containing 1.0 or 0.5 g. Product made of cocoa bean fibers and oat fibers. Usage ad libitum. Recommended dosages: 10-24 sachets per day (1.0 g sachets). Among participants who typically smoke >15-20 cigarettes per day and/or has a Fagerström score of 7 or higher, the recommended maximum number of sachets per day is 30. For participants who use small sachets (0.5 g) the recommended daily use is double compared that of 1.0 g sachets.
  Arms: 2

SUMMARY:
The study aims to assess if use of a low-nitrosamine, Swedish, smokefree tobacco product for oral use ("snus") can increase the quit rate among cigarette smokers who wish to stop smoking

DETAILED DESCRIPTION:
In a multicenter, double-blind, placebo-controlled setting, participants are randomly allocated to either a smokefree, oral tobacco product or a non-tobacco, non-nicotine placebo product with identical flavoring and physical appearance. The study consists of three phases: Study Product Test Period (4 weeks), Intervention Phase (12 weeks), and a Follow-Up Phase (12 weeks). The participants are all cigarette smokers who are motivated to quit. They are encouraged to gradually substitute as many cigarettes as possible with study products during the Study Product Test Period and to refrain from all cigarettes at the latest by the first day of Week 5. Use of study products will continue during the 12 week Intervention Phase. The participants are encouraged to cut down on use of study products during the last 3 weeks to avoid a too abrupt ending of nicotine intake.

All subjects are encouraged to continue in the study for clinical follow-up independent of smoking status although use of study products is discontinued during the Follow-Up Phase. If a subject has managed to quit smoking during the Intervention Phase but there is an imminent danger of smoking relapse during the Follow-Up Phase, that subject is informed that use of nicotine replacement therapy or a smokefree tobacco product is a better option in terms of health risks than a smoking relapse.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smoker who smoke more than 9 cigarettes per day (average during past month)
* Daily smoking more than 1 year
* Motivated to quit smoking using a smokefree tobacco product
* Good general health

Exclusion Criteria:

* Use of smokefree/smokeless tobacco during past 6 months or any type of pharmaceutical product for smoking cessation during past 3 months
* Unable to refrain from nicotine replacement therapy during the study
* Current oral condition that could be made worse by study interventions
* History of clinically significant renal, hepatic, neurological, or chronic pulmonary disease that in the judgement of the investigator might preclude participation
* History of significant cardiovascular disease, including myocardial infarction, within the last 3 months, significant cardiac arrythmias, or poorly controlled hypertension that in the judgement of the investigator might preclude participation
* History of alcohol or substance abuse other than cigarette smoking within the past year

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Fagerström, Ph. D., Study Chair — Smoker's Information Center, Hälsingborg, Sweden; Randall R Stoltz, MD, Principal Investigator — Covance Clinical Research Unit, Evansville, In; Frank H Farmer, Jr, MD, Ph D, CPI, Principal Investigator — Covance Clinical Research Unit, Daytona Beach, FL; David C Carter, MD, Principal Investigator — Covance Clinical Research Unit, Austin, TX; Keith Klatt, MD, Principal Investigator — Covance Clinical Research Unit, Portland, OR
Locations (4):
- United States (4):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Evansville, Indiana
  - Covance Clinical Research Unit, Portland, Oregon
  - Covance Clinical Research Unit, Austin, Texas

REFERENCES:
- [Result] Fagerstrom K, Rutqvist LE, Hughes JR. Snus as a smoking cessation aid: a randomized placebo-controlled trial. Nicotine Tob Res. 2012 Mar;14(3):306-12. doi: 10.1093/ntr/ntr214. Epub 2011 Oct 12. PMID 21994343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from database of clinical trial volunteers, and media ads
Pre-assignment Details: Participants were checked for eligibility prior to group assignment
Groups:
- Active Snus: Tobacco-based, smokefree product
- Placebo Snus: Non-tobacco, non-nicotine placebo product
Period: Overall Study
Arm/Group | Active Snus | Placebo Snus
Started | 125 | 125
Completed | 82 | 70
Not Completed | 43 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Snus | Placebo Snus | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 125 | 250
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 71 | 152
  Male | 44 | 54 | 98
Region of Enrollment [Number; unit: participants]
  United States | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Continuous Rate of Smoking Cessation by Self-report and Confirmed by Expired Air Carbon Monoxide Less or Equal Than 8 Ppm
Time Frame: Week 6-28
Measure: Number; unit: participants
Arm/Group | Active Snus | Placebo Snus
Number analyzed (Participants) | 125 | 125
participants | 5 | 2

2. Secondary Outcome: Minnesota Nicotine Withdrawal Scale
Time Frame: Baseline, week 6, 10, 16 and 28
Reporting Status: Not Posted

3. Secondary Outcome: Fagerström Test for Nicotine Dependence
Time Frame: Baseline, week 16 and 28
Reporting Status: Not Posted

4. Secondary Outcome: Biomarkers
Time Frame: Baseline, week 6, 16, and 28
Reporting Status: Not Posted

5. Secondary Outcome: Point Prevalence Smoking Cessation
Description: 7-day point prevalence smoking cessation verified by CO in exhaled air of 8 ppm or less
Time Frame: 6, 16, 28 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Continuous Smoking Cessation
Description: Continuous cessation according to self-report and CO in exhaled air of 8 ppm or less att all clinical visits
Time Frame: 6-16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Active Snus | Placebo Snus
Serious Adverse Events (participants affected / at risk) | 2/125 | 2/125
Other Adverse Events (participants affected / at risk) | 53/125 | 37/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Snus (N=125) | Placebo Snus (N=125)
Vaginal bleeding (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Severe visual disturbance (Nervous system disorders) | 0 | 1 (1) — Severe visual disturbance secondary to cerebrovascular incident
severe multiple fractures in right ankle due to car accident (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Snus (N=125) | Placebo Snus (N=125)
Gingival pain, nausea, dyspepsia etc (Gastrointestinal disorders) | 53 (53) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No